CLINICAL TRIAL: NCT03847467
Title: Pilot and Feasibility Study of 2'-FL as a Dietary Supplement in Pediatric and Young Adult IBD Patients Receiving Stable Maintenance Anti-TNF Therapy
Brief Title: Pilot and Feasibility Study of 2'-FL as a Dietary Supplement in IBD Patients Receiving Stable Maintenance Anti-TNF Therapy
Acronym: PRIME
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Broad Institute of MIT and Harvard (Other); University of Cincinnati (Other); Connecticut Children's Medical Center (Other); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-6667
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — 2'-fucosyllactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2'-Fucosyllactose (Experimental): Phase I: 36 young adult participants aged 18-25 years. Group 1: 1 gm per day n=12 (6UC/6CD) Group 2: 5 gm per day n=12 (6UC/6CD) Group 3: 10 gm per day n=12 (6UC/6CD)
  Phase II (post Phase I interim safety analysis): 120 participants aged 11-25 years Group 1: 1 gm per day n=40 (20UC/20CD) Group 2: 5 gm per day n=40 (20UC/20CD) Group 3: 10 gm per day n=40 (20UC/20CD)
  Interventions: Drug: 2'-Fucosyllactose
- Placebo (Placebo Comparator): Phase I: 20 young adult participants age 18-25 years dosed at 2 gm placebo per day. (10UC/10CD)
  Phase II (post Phase I interim safety analysis): 40 participants age 11-25 years dosed at 2 gm placebo per day. (20UC/20CD)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2'-Fucosyllactose — Human milk oligosaccharide prebiotic dietary supplement
  Other Names: 2'-FL
  Arms: 2'-Fucosyllactose
Other: Placebo — Dextrose
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled dose-ranging study of 2'-FL in IBD, Crohn's Disease (CD) and ulcerative colitis (UC). The overarching hypothesis is that 2'-FL supplementation in IBD will be safe and well tolerated, while increasing fecal Bifidobacterium abundance and butyrate in a dose dependent manner. The investigators will test 1, 5, or 10 gm 2'-FL compared to 2 gm dextrose placebo as a daily dietary supplement in pediatric and young adult IBD participants in stable remission receiving infliximab, adalimumab, or infliximab-dyyb biosimilar anti-TNF therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 11 - 25
4. Diagnosed with Crohns Disease or Ulcerative Colitis
5. Disease is in remission

   * Adult CD (age 18-25): CDAI score < 150
   * Pediatric CD (age 11-17): wPCDAI < 12.5
   * Adult UC (age 18-25): Modified Mayo sub-scores: stool frequency sub-score=0, rectal bleeding sub-score=0
   * Pediatric UC (age 11-17): PUCAI score < 10
6. Not receiving corticosteroids
7. Receiving a stable anti-TNF maintenance dose of adalimumab, infliximab, or the biosimilar infliximab-dyyb for 12 weeks prior to enrollment. A stable infliximab or infliximab-dyyb dose may range from 5 mg/kg every 8 weeks to 10 mg/kg every 4 weeks. A stable adalimumab dose may range from 20 mg every 2 weeks to 40 mg every 7 days. While therapeutic drug monitoring will not be required for inclusion, all drug and anti-drug antibody levels obtained for clinical indications within six months prior to enrollment, and from the screening visit through week 20, will be recorded.
8. If receiving mesalamine, mercaptopurine, azathioprine, or methotrexate, must be on a stable dose for at least 12 weeks prior to enrollment.
9. Agreement to not make any major dietary changes throughout study duration. This would include changing usual diet to a vegan diet, Specific Carbohydrate Diet (SCD), or exclusive enteral nutrition (EEN) diet.
10. We will include CD patients who have had one ileo-colic resection, as long as the resection did not include more of the colon than the cecum and ascending colon. CD patients may be enrolled if at least six months post-surgery.

Exclusion Criteria:

1. Experienced active IBD clinical disease during the previous six months as determined by the Principal Investigator.
2. Use of any of the following medications during the previous month: antibiotics, probiotics or prebiotics
3. Diagnosis of celiac disease, diabetes or other co-morbidity that is determined by the PI as being exclusionary
4. Treatment with another investigational drug or other intervention within 4 weeks
5. Treatment with other biologic medication for IBD within prior 12 weeks
6. Problem with lactose breakdown
7. Currently pregnant or breast feeding
8. We will exclude CD patients with more than one IBD related surgery, or those with a sub-total colectomy. We will exclude UC patients with colectomy or IBD related surgery.
9. We will not allow concomitant use of anti-diarrheal medications.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Gastrointestinal Symptom Rating Scale (GSRS) in participants who receive 2'-fucosyllactose (2'FL) or dextrose placebo | 20 weeks
  Measured by the Gastrointestinal Symptom Rating Scale (GSRS). The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire for patients with GI symptoms. Patients are asked to numerically score their subjective symptoms on a scale of 1-7 (1=no discomfort up to 7=severe discomfort). The sum of the scores for all 15 items is regarded as the GSRS total score

SECONDARY OUTCOMES:
Mean fecal Bifidobacterium abundance in participants who receive 2'-fucosyllactose (2'FL) or dextrose placebo | 20 weeks
  Measured by fecal DNA 16S ribosomal sequencing

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No